CLINICAL TRIAL: NCT00676754
Title: Epidemiology of Multidrug-Resistant Tuberculosis in Peru
Brief Title: Epidemiology of MDR-TB in Peru
Acronym: Estudio Epi
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Harvard University Faculty of Medicine (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other); Brigham and Women's Hospital (Other); Socios En Salud Sucursal, Peru (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Mercedes Becerra, Associate Professor of Global Health and Social Medicine, Harvard University Faculty of Medicine
Other Study IDs: 07-0002; 5U19AI076217 (NIH); R01AI057786 (NIH)
Record Dates: First submitted 2008-05-08; First posted 2008-05-13 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: TB Multi-drug Resistant
Keywords: Multidrug-Resistant Tuberculosis, tuberculosis, Peru
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant; Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, sputum
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Statens Serum Institut RT23 2TU tuberculin

SUMMARY:
The purpose of this study is to better understand tuberculosis (TB) and the risk of infection with TB, in Peru. TB is a disease that is caused by bacteria and transmitted through droplets in the air that come from the lungs of an infected person. The risk of infection will be compared between two groups: household members, who live with people having TB that does not respond well to treatment and household members, who live with people having TB that responds well to treatment. Study participants will include 4,500 TB infected people and 22,500 of their household contacts. Study procedures include answering a questionnaire, TB skin tests, blood samples, and a chest x-ray. Individuals with symptoms indicating TB will be asked to provide sputum samples. Individuals with TB will be involved in the study for up to 48 months; household contacts will be involved in the study for 12 months. The knowledge gained from this study will be used to improve tuberculosis control.

DETAILED DESCRIPTION:
The emergence of drug-resistant and multi-drug resistant Mycobacterium (M) tuberculosis poses a significant threat to global tuberculosis (TB) control strategies. The prospective design of this study will allow the direct study of infection risk, because the population among which the TB cases arise will be identified and monitored over the course of the study. This study design will permit the characterization and comparison of TB strains with differential success in causing new infections. The study will be conducted within a well-established public health TB control program in a region of Peru, where drug-resistant strains already account for about 20 percent of new TB cases. This study protocol will be implemented in collaboration with the 52 Ministry of Health outpatient health centers in 4 districts of Lima, Peru. This will be a prospective cohort study with an enrollment period of 36 consecutive months. Two types of study subjects will be enrolled: patients found to have active TB disease by routine testing (TB index subjects), and the individuals living in the households of these patients (household members). Study participants will include 4,500 subjects with active TB and their approximately 22,500 household members. Ages will range from less than 1-100 years. The tuberculin skin test will be used to diagnose latent TB infection in the household members. This product is used routinely by health center staff in household members who are children in the age group less than1-15 years. In this study protocol, it will also be used in all household members age 16 years and older. Each TB index subject will remain in the study for a minimum of 12 months and a maximum 48 months. Each household member will remain in the study for 12 months. The primary objective of the study is to measure the risk of infection in household members of index cases with drug-resistant TB compared with the risk of infection in household members of subjects with drug-sensitive TB. This refers to household members who are tuberculin-skin-test negative at the beginning of follow-up. Secondary study objectives are: to assess the impact of sociodemographic and clinical confounders and risk modifiers such as age, sex, comorbidity, human immunodeficiency virus (HIV) infection, nutritional status, and Bacille Calmette Guerin (BCG) vaccination on the association between risk of infection and exposure to a drug-resistant or a drug-sensitive strain; to measure associations between specific mutations associated with drug resistance in M tuberculosis and phenotypes including resistance profile, clinical presentations, and transmissibility; to measure the rate of true relapse versus reinfection in drug-resistant and drug-sensitive TB subjects using molecular-epidemiologic methods; and to measure the rate of reversion (to negative) of the tuberculin skin test among household members with a positive tuberculin skin test result. The primary study outcome measure is the relative risk of TB infection (by tuberculin skin test) in household members of subjects who are sick with drug-resistant M tuberculosis strains compared to household members of subjects with drug-sensitive strains. Secondary study outcome measures are the rate of relapse and rate of reinfection among TB subjects treated with routine TB therapy by outpatient health centers; and the rate of reversion (to negative) of the tuberculin skin test among household members with a positive tuberculin skin test result.

ELIGIBILITY:
Inclusion Criteria:

TB index subjects

* During the enrollment period, the participant is found to have characteristic acid-fast bacilli shown by the Ziehl-Neelsen stain on a smear of sputum indicating active disease due to M. tuberculosis.
* Participant is at least 16 years old at the time of enrollment.
* Participant lives in one of the study districts.
* If age 18 years or older, participant provides informed consent to participate. If age 16 or 17 years, a guardian provides informed consent for minor to participate, and the minor also provides assent.

Household members

* Participant lives in the same household as an index subject at the time the index subject is enrolled in the study.
* If eligible participant is age 18 years or older, participant provides informed consent to participate. If participant is younger than 18 years, a parent or guardian provides informed consent for minor to participate. If eligible participant is age 10-17 years, the minor also provides assent.

Exclusion Criteria:

* Apart from the age restriction (age 16 years and older) for the group of TB index subjects, no other exclusion criteria apply.
* Previous diagnosis with TB disease will not be considered a reason for exclusion from the study.
* Pregnant or breast-feeding women will be eligible to participate in the study.
* Prior to beginning routine TB treatment, health center workers provide women with routine counseling about the use of contraceptive methods during TB treatment; this is not a study activity.
* Subjects who live alone will be included in the study and will contribute to addressing the third and fourth study objectives.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes two categories of subjects: (1) the 4,000 TB index subjects and (2) their approximately 18,000 household members. All of these individuals live in Lima, Peru, in the catchment area of the participating public health centers.
  Approximately 50% of study participants will be female. According to the ethnic and racial categories used by NIH, all of the study population would be classified as "Hispanic or Latino" (Mestizo). None of these participants live within a tribal indigenous culture; all speak Spanish while some also speak the indigenous (Quechua) language of their birthplace in Peru. At least 75% of this population has some "Amerindian" heritage. Less than 1% of individuals are either Asian-Peruvian or Afro-Peruvian in descent.
  Apart from the age restriction (at least 16 years old) for the TB index subjects only, there are no other restrictions on participant selection
Sampling Method: Non-Probability Sample
Enrollment: 18544 (Actual)
Dates: Start 2009-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Risk of TB infection among the household members | at months 6 and 12 after study enrollment

SECONDARY OUTCOMES:
Relative risk of specific DR mutations in index case across household contacts who acquire TB from strain matching the index case strain, vs. disease-free contacts; and cases whose contacts do/do not convert from negative to positive PPD skin test. | at months 6 and 12 after study enrollment

OTHER OUTCOMES:
Relative risk of relapse and reinfection in index patients who are sick with drug-resistant M. tuberculosis strains compared to index patients sick with drug-sensitive strains. | 24-month period after completing TB drug therapy

CONTACTS AND LOCATIONS:
Overall Officials: Megan Murray, MD, ScD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (1):
- Socios En Salud Sucursal Peru, Lima, Peru

REFERENCES:
- [Derived] Becerra MC, Huang CC, Lecca L, Bayona J, Contreras C, Calderon R, Yataco R, Galea J, Zhang Z, Atwood S, Cohen T, Mitnick CD, Farmer P, Murray M. Transmissibility and potential for disease progression of drug resistant Mycobacterium tuberculosis: prospective cohort study. BMJ. 2019 Oct 24;367:l5894. doi: 10.1136/bmj.l5894. PMID 31649017